CLINICAL TRIAL: NCT03677102
Title: Fluids in Septic Shock (FISSH): a Randomized Controlled Trial
Brief Title: Fluids in Septic Shock (FISSH)
Acronym: FISSH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1515
Record Dates: First submitted 2018-08-27; First posted 2018-09-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sepsis, Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- higher chloride solutions (Active Comparator): higher chloride crystalloid (Normal saline - chloride concentration 154 mmol/L)
  Interventions: Other: higher chloride crystalloid
- lower chloride solutions (Active Comparator): lower chloride crystalloid (Ringer's lactate - chloride concentration 110 mmol/L)
  Interventions: Other: lower chloride crystalloid

INTERVENTIONS:
Other: higher chloride crystalloid — Normal saline (chloride concentration 154 mmol/L)
  Arms: higher chloride solutions
Other: lower chloride crystalloid — Ringer's Lactate (chloride concentration 110 mmol/L)
  Arms: lower chloride solutions

SUMMARY:
Despite evidence of the physiologic benefits and possible lower mortality associated with low chloride solutions, normal saline remains the most wildly used fluid in the world. Given uncertainty about the impact of lower chloride versus higher chloride solutions on mortality, it is unlikely that clinical practice will change without new and direct randomized controlled trial (RCT) evidence. Editorials published in leading critical care journals have called for RCT's to address this important clinical question. This trial will directly compare low chloride versus normal chloride for resuscitation in septic shock on patient-important outcomes such as mortality and AKI.

DETAILED DESCRIPTION:
Severe infection can lead to many complications within the human body including low blood pressure, which is called septic shock. The main treatments for septic shock are intravenous antibiotics and intravenous fluid.

There are many different intravenous fluids available for doctors to use. Each one of these fluids has potential advantages as well as potential disadvantages. Doctors will often look at many things when deciding which fluid to give including the results of bloodwork and the clinical characteristics of the patients themselves. There is limited direction from research studies that using one fluid type is better than another. Some preliminary research in the field has suggested that one specific electrolyte, call chloride, may be harmful when given to patients in high concentrations. Animal research has shown that the administration of high chloride fluids may be harmful to the lungs, kidneys, gastrointestinal and muscle cells. Some intravenous fluids have higher concentrations of chloride than others.

The investigators plan to study the impact of giving patients with severe infection intravenous fluids with either a high chloride concentration (normal saline or high chloride albumin) or a low chloride concentration (Ringers Lactate or low chloride albumin). This trial will build on the earlier pilot, phase 1 study and will look at patient-important outcomes such as rate of death, kidney failure and length of stay in the ICU. This larger study has the potential to guide the care of critically ill patients with infection worldwide.

ELIGIBILITY:
Inclusion Criteria:

* patients 16 years or greater who meet all of the following:
* require fluid resuscitation for refractory hypotension (systolic blood pressure <90 mmHg or mean arterial blood pressure<65 mmHg after 1 Litre bolus over 1 hour or less or organ hypo-perfusion (serum lactate >4 mmol/L)
* have a clinical suspicion of infection
* are within 6 hours of hospital admission or critical care response team consultation
* are anticipated to require ICU admission

Exclusion Criteria:

* intracranial bleed or intracranial hypertension during the index hospital admission
* 10% of body surface area acute burn injury
* bleeding/hemorrhage as likely cause of hypotension
* a lack of commitment to life support
* have previously enrolled in FISSH, or a confounding trial (e.g. a trial examining the effect of other intravenous fluids in septic shock patients)
* been transferred from another hospital or facility >6 hours since presentation to first hospital
* pre-established end stage renal disease (ESRD) or are receiving hemodialysis (intermittent or continuous) at time of enrolment, or
* been admitted to ICU directly from the operating room or post anaesthetic care unit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1096 (Estimated)
Dates: Start 2018-09-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
30-day Mortality | up to 30 days
  We expect that if a difference in survival is demonstrated, that this will be evident within 30 days

SECONDARY OUTCOMES:
Acute Kidney Injury | up to 30 days
  Development of stage 2 or worse acute kidney injury (AKI) according to KIDGO guidelines on serum creatinine criteria

OTHER OUTCOMES:
Hospital/ICU length of stay | up to 30 days
  length of hospital/ICU stay up to 30 days
Ventilator free days | censored at 30 days
  Number of ventilator free days
Number of days requiring vasoactive agents | up to 30 days
  defined as the number of days requiring great than or equal to 2 hours of intravenous vasopressor support
Incidence of biochemical abnormalities during study period | up to 30 days
  any serum blood test results showing hyperchloremia, hyperkalemia, hypernatremia, or acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Bram Rochwerg, MSc,MD,FRCPC, Principal Investigator — McMaster University
Locations (29):
- Canada (27):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Calgary - Rockyview General Hospital, Calgary, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Halifax Infirmary, Halifax, Nova Scotia
  - Victoria General, Halifax, Nova Scotia
  - Cape Breton Regional Hospital, Sydney, Nova Scotia
  - Lakeridge Health - Ajax Pickering, Ajax, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - St Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Hospital-Hamilton Health Sciences, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - London Health Sciences - University Hospital, London, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Niagara Health, St Catharines Site, St. Catharines, Ontario
  - Unity Health (St. Michael's Hospital), Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Hospital - Ouellette Campus, Windsor, Ontario
  - Windsor Regional Hospital -Metropolitan Campus, Windsor, Ontario
  - Centre intégré Universitaire de santé et de services sociaux du Nord de l'île de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Centre de recherche du CIUSSS de l'Estrie - CHUS de Sherbrooke, Sherbrooke, Quebec
  - Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec (CIUSSS MCQ), Trois-Rivières, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - St Paul's Hospital, Saskatoon, Saskatchewan
- Saudi Arabia (2):
  - King Abdulaziz Medical City- Riyadh (KAMC-R), Riyadh
  - King Faisal Specialist Hospital & Research Centre, Riyadh

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03677102/Prot_SAP_000.pdf